CLINICAL TRIAL: NCT06101108
Title: Early Diagnosis of Age-Linked CArdiac TransThyRetin Amyloidosis by Selective Screening in Spinal Stenosis Surgery: the Multi-centric ALCATTRASS-study.
Brief Title: Early Diagnosis of Age-Linked CArdiac TransThyRetin Amyloidosis by Selective Screening in Spinal Stenosis Surgery
Acronym: ALCATTRASS
Status: Recruiting | Type: Observational
Sponsor: Philippe Debonnaire (Other)
Responsible Party: Sponsor-Investigator, Philippe Debonnaire, Chief Investigator, AZ Sint-Jan AV
Organization: AZ Sint-Jan AV (Other)
Other Study IDs: ALCATTRASS
Record Dates: First submitted 2023-10-20; First posted 2023-10-26 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Transthyretin Amyloid Cardiomyopathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to keep track of the cardiological follow-up of patients who have undergone back surgery because of symptomatic narrowing of the spinal canal and in whom microscopic examination of the tissue removed during this surgery showed a high amount of local deposits of small proteins. This finding may be an early sign of a condition in which other organs (especially the heart) may also be affected by these proteins, called amyloidosis.

Patients who participate in this study, will be followed up for life. During the first routine consultation with the cardiologist, the physician-investigator will collect information, such as demographics (age, weight, height, gender), medical history, medication, symptoms and the results of prescribed examinations. These examinations include microscopic examination of tissue removed during the surgery, blood tests, electrocardiography, echocardiography and a bone scan. These examinations are clinically necessary and appropriate, and patients should undergo them even without participating in the study.

DETAILED DESCRIPTION:
Background: Transthyretin amyloid cardiomyopathy (ATTR-CM) is an underdiagnosed, severe, yet treatable disease. Lumbar spinal stenosis (SS) in elderly is a red flag for ATTR-CM, often preceding cardiac diagnose by many years. Yet, optimal screening strategies for early ATTR-CM detection at time of SS diagnosis are underused.

Study aim: Multi-centric validation of the diagnostic yield of a standard-of-care prospective screening strategy for early ATTR-CM detection in the elderly, based on ligamentum flavum biopsy assessment at SS surgery.

Design: International, multi-centre, prospective, observational, multi-disciplinary, diagnostic registry.

Methods: All consecutive patients ≥60 years old undergoing standard-of-care ligamentum flavum biopsy as part of symptomatic SS surgery within 12 heart centres are included. The burden of ATTR amyloid deposition (positive Congo-red and pre-albumin staining) is assessed semi-quantitatively by visual Westermark grading. Patients with significant ATTR amyloid burden (grade 3 (≥5-10%) or 4 (>10%) ATTR amyloid on biopsy specimen) undergo standard-of-care work-up to exclude ATTR-CM, conform state-of-the-art clinical practice and ESC recommendations (i.e. baseline cardiac biomarkers, ECG, transthoracic echocardiography, monoclonality assessment and bone-scintigraphy with SPECT; additional CMR and/or endomyocardial biopsy as needed). The diagnostic yield of this biopsy-based strategy will be evaluated.

Conclusion: This trial will validate the diagnostic yield of selective ligamentum flavum biopsy analysis in SS surgery patients as a simple and valuable prospective screening strategy for early ATTR-CM detection.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 60 years old
* Lumbar spinal canal stenosis, undergoing spinal surgery
* Westermark grade 3 or 4 ATTR amyloid burden on ligamentum flavum biopsy

Exclusion Criteria:

* Prior diagnosis of cardiac amyloidosis
* Unwilling to provide informed consent

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive patients ≥60 years old that undergo lumbar spinal stenosis surgery at the neurosurgery or orthopaedic department with Westermark grade 3 or 4 ATTR amyloid burden on ligamentum flavum biopsy
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2024-06-24 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Rate of diagnosis of cardiac amyloidosis | 1 week
  Diagnosis of transthyretin amyloid cardiomyopathy

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Debonnaire, MD, PhD, Principal Investigator — AZ Sint-Jan Brugge AV
Locations (1):
- AZ Sint-Jan Brugge AV, Bruges, Belgium

IPD SHARING:
Plan to Share IPD: No